CLINICAL TRIAL: NCT03211442
Title: Implications of MEDIcal Low Dose RADiation Exposure - BReast Cancer Acute Coronary Events (MEDIRAD-BRACE): A Retrospective Cohort Study
Brief Title: Implications of MEDIcal Low Dose RADiation Exposure - BReast Cancer Acute Coronary Events
Acronym: MEDIRAD-BRACE
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: The Netherlands Cancer Institute (Other); Technical University of Munich (Other); Institut de Radioprotection et de Surete Nucleaire (Other Government)
Responsible Party: Sponsor
Other Study IDs: RT2017-08
Record Dates: First submitted 2017-07-06; First posted 2017-07-07 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer Female; Acute Coronary Events; Cardiac Complications
Keywords: Breast cancer; Radiotherapy; Cardiac complications; Acute coronary events; NTCP model
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radiotherapy — Breast cancer patients treated with radiotherapy

SUMMARY:
MEDIRAD-BRACE aims to determine the relationship between 3D dose distributions in cardiac structures and the risk of acute coronary events (ACE) and other cardiac complications in breast cancer (BC) patients to develop and externally validate multivariable Normal Tissue Complication Probability (NTCP) models to assess the risk of ACE in individual patients based on cardiac dose metrics in the first 10 years after BC radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients;
* Treated with primary surgery for stage I-III invasive adenocarcinoma of the breast or ductal carcinoma in situ (DCIS);
* Age between 40-75 years at time of start RT;
* WHO performance status 0-1;
* Planned for RT alone to the breast, the chest wall and/or the lymph node areas;
* Start of RT is between 01-01-2015 and 31-12-2013;
* Available planning CT scan and dose distribution;
* Adjuvant systemic treatment, including hormonal therapy or chemotherapy is allowed;
* Medical history of coronary artery disease and/or myocardial infarction is not an exclusion criterion;
* Written informed consent.

Exclusion Criteria:

* Male breast cancer patients;
* Women with metastatic breast cancer (M1 disease);
* Any prior malignancy other than non-melanoma skin cancer;
* Previous thoracic or mediastinal radiation;
* Women treated with neoadjuvant chemotherapy.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, female patients with stage I-III breast cancer, treated with primary surgery, either by mastectomy of breast conserving surgery, and postoperative RT in the period 2005-2013, and who were aged 40-75 years at the time of RT
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with an Acute Coronary Event after completion of RT treatment | First 10 years after RT treatment

SECONDARY OUTCOMES:
Number of patients with other cardiac complications after completion of RT treatment | First 10 years after RT treatment
Number of patients with radiotherapy-induced late non-cardiac toxicity (e.g. secondary tumors) | First 10 years after RT treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Errahmani MY, Locquet M, Spoor D, Jimenez G, Camilleri J, Bernier MO, Broggio D, Monceau V, Ferrieres J, Thariat J, Boveda S, Kirova Y, Loap P, Langendijk JA, Crijns A, Jacob S. Association Between Cardiac Radiation Exposure and the Risk of Arrhythmia in Breast Cancer Patients Treated With Radiotherapy: A Case-Control Study. Front Oncol. 2022 Jul 4;12:892882. doi: 10.3389/fonc.2022.892882. eCollection 2022. PMID 35860581